CLINICAL TRIAL: NCT05635175
Title: Effectiveness of a Hip Abductor Training in Women With Stress Urinary Incontinence
Acronym: PROTOGLUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: GIRCI NO (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/0176/HP
Record Dates: First submitted 2022-11-03; First posted 2022-12-02 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Women With Stress Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physiotherapist-supervised pelvic floor muscle training (Active Comparator): physiotherapist-supervised pelvic floor muscle (PFM) training (PFMT) and self training PFMT
  Interventions: Other: Standard pelvic floor muscle training; Other: Standard pelvic floor muscle training self training
- hip abductors self training program (Experimental): physiotherapist-supervised pelvic floor muscle (PFM) training (PFMT) and self training hip abductors self training program
  Interventions: Other: hip abductors physiotherapy self training; Other: Standard pelvic floor muscle training

INTERVENTIONS:
Other: hip abductors physiotherapy self training — hip abductors self training program during 7 to 10 weeks associate with a PFMT
  Arms: hip abductors self training program
Other: Standard pelvic floor muscle training — Standard pelvic floor muscle training
Other: Standard pelvic floor muscle training self training — Standard pelvic floor muscle training self training
  Arms: physiotherapist-supervised pelvic floor muscle training

SUMMARY:
Urinary incontinence (UI) is estimated to affect 25% à 45 % women all over the world. UI is associated with a poor Quality of life, with a strong level of certainty. Stress urinary incontinence (SUI) is the second more prevalent type of UI . First-line treatment for SUI is conservative, non-drug and non-surgical treatment. Among these techniques, physiotherapist-supervised pelvic floor muscle (PFM) training (PFMT) as a first-line treatment; however, only half of women with SUI are cured with PFMT.

Brain imaging shows that PFMs (involved in continence mechanisms) and gluteal muscles can activate the same cortical region. This synergy is found if the gluteal muscles are voluntarily activated, but not if the PFMs are volontary activated alone . In women, hip abductor physiotherapy is a common practice which has already been the subject of a very extensive literature and has largely shown its effectiveness in the quality of lumbo-pelvic control, balance, quality of life and risk of fall prevention. This rehabilitation is based on exercises that induce solicitation of the hip abductors by synergistic reflex activation during a range of well-known exercises. Recent work has shown the effect of hip abductors on the activation of the PFMs . Until today, there is no literature evaluating the effectiveness of a hip abductors training program without associated voluntary contraction of the PFMs (PPM) on UI. The hypothesis of this work will be to demonstrate that a complementary training focused on the hip abductor, complementary to concomitant PFMT, would benefit from a more significant improvement in continence, and also in physical abilities and quality of life. Because balance seems involved in UI, we therefore propose to to observe the effects on the frontal balance of the pelvis. As the investigators have already done in previous studies, to identifying factors that predict the success of our interventions, investiagtors have planned to evaluate the observance and adherence of our patients .Complementary, the investigators planned to evaluate the effect of both intervention on pelvic floor muscles and hip abductors strength and endurance, pelvic organ prolapse symptoms and quality of life. For this objective, the investigators intend to compare two randomized parallel groups: Group A follow a 12 sessions supervised PFMT + home based PFMs exercices. Group B follow a 12 sessions supervised PFMT + home based hip abductor exercices.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 ans
* patient with urinary incontinence according to the ICS criteria [3]
* having received a prescription for perineal rehabilitation
* affiliated to french health care insurance
* Patient having read and understood the information letter and signed the consent form
* Effective contraception in women of childbearing age (negative urine pregnancy test). For postmenopausal women, a confirmatory diagnosis must be obtained (amenorrhea for at least 12 months before the inclusion visit)

Exclusion Criteria:

* Bladder pathologies (cyst, tumour, interstitial cystitis)
* Neurological pathologies (multiple sclerosis, Parkinson's desease, etc.)
* Pregnant or parturient or breastfeeding woman or absence of proven contraception
* Person deprived of liberty by administrative or judicial decision or a person placed under the safeguard of justice, or guardianship or curatorship
* Physical inability to perform hip abductors exercises (unable to walk or stand independently)
* Women having scheduled continence surgery before the end of physiotherapy sessions at the time of randomization
* Women having at least one of the continence-specific anticholinergic treatments prescribed before the end of the physiotherapy sessions at the time of randomization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-23 (Estimated)

PRIMARY OUTCOMES:
The difference in the number of leaks per week observed after the end of treatment between the two arms at the last physiotherapy session. | 10 weeks
  This number of leaks per week will be recorded using question 3 of the International Consultation on Incontinence Questionnaire (ICIQ-SF).

SECONDARY OUTCOMES:
Measurement in centimeters of the offset in the frontal plane of the postero-superior iliac spines during a one leg stance | 10 weeks
Average of the measurement in Newton of the force of the hip abductors during a maximum manual resistance test repeated 3 times using a dynamometer | 10 weeks
Average of measurement in seconds of the hip abductors resistance during a manual resistance test repeated 10 times | 10 weeks
Measurement rated from 1 to 5 of the strength of PFMs according to the "Modified Oxford Grading Scale" testing | 10 weeks
Overall score and sub-scores of urinary symptoms from the international consultation on incontinence questionnaire | 10 weeks
  min: 0 : better outcome max : 21 worse outcome
Overall score and sub-scores of urinary symptoms of the Prolape quality of life questionnaire | 10 weeks
Short Form-36 Quality of Life overall score and subscores | 10 weeks
Overall score and sub-scores of physical inactivity and physical abilities from the Ricci & Gagnon questionnaire | 10 weeks
Overall score and sub-scores of the therapeutic observance and adherence questionnaire (only at the end of treatment) | 10 weeks
Patient Global Impression of Improvement (PGI-I) questionnaire score (only at end of treatment) | 10 weeks
Overall score and sub-scores of urinary symptoms from the international consultation on incontinence questionnaire questionnaire | through study completion, an average of 6 month
Overall score and sub-scores of urinary symptoms of the Prolapsus Quality of Life questionnaire 3. SF-36 Quality of Life overall score and subscores | throught study completion, an average of 6 month
Overall score and sub-scores of physical inactivity and physical abilities from the Ricci & Gagnon questionnaire | throught study completion, an average of 6 month
Score du questionnaire Patient Global Impression of Improvement (PGI-I) | throught study completion, an average of 6 month
  min: 1 better outcome max : 7 worse outcome

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Pôle santé de la Grace Dieu, Caen
  - Chu Rouen, Rouen
  - Médipôle du Rouvray, Saint-Étienne-du-Rouvray

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stewart WF, Hirsh AG, Kirchner HL, Clarke DN, Litchtenfeld MJ, Minassian VA. Urinary incontinence incidence: quantitative meta-analysis of factors that explain variation. J Urol. 2014 Apr;191(4):996-1002. doi: 10.1016/j.juro.2013.10.050. Epub 2013 Oct 16. PMID 24140547
- [Background] Ebbesen MH, Hunskaar S, Rortveit G, Hannestad YS. Prevalence, incidence and remission of urinary incontinence in women: longitudinal data from the Norwegian HUNT study (EPINCONT). BMC Urol. 2013 May 30;13:27. doi: 10.1186/1471-2490-13-27. PMID 23721491
- [Background] Pizzol D, Demurtas J, Celotto S, Maggi S, Smith L, Angiolelli G, Trott M, Yang L, Veronese N. Urinary incontinence and quality of life: a systematic review and meta-analysis. Aging Clin Exp Res. 2021 Jan;33(1):25-35. doi: 10.1007/s40520-020-01712-y. Epub 2020 Sep 22. PMID 32964401
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322
- See also: Steenstrup B, M. Pavy Lebrun, Aigueperse N, Quemener N, Cheveau S, Confalonieri C, Totte F. Efficacité d'une rééducation sensori-motrice posturale réflexe sur l'incontinence urinaire et l'urgenturie chez la femme. Kinesith Rev. 2019;19(206):12-18 — https://doi.org/10.1016/j.kine.2018.11.005
- See also: Steenstrup B, Behague L, Quehen M. Rééducation posturale avec le jeu virtuel Wii ® en pelvi périnéologie: pourquoi pas? Kinésith Rev. 2015;15(160):45-50 — https://doi.org/10.1016/j.kine.2014.11.087